CLINICAL TRIAL: NCT06012643
Title: Subperiosteal Implants as a Treatment for Severely Atrophied Jaw in Completely and Partially Edentulous Population: A Systematic Review of Case Reports and Case Series.
Brief Title: Subperiosteal Implants Constructed With Digital Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Elsawy, lecturer, Department of prosthodontics, principle investigator, Mansoura University
Other Study IDs: A0107023RP
Record Dates: First submitted 2023-08-13; First posted 2023-08-25 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The purpose of this systematic review of case reports and case series was to evaluate the spectrum of subperiosteal implants for severely atrophied jaws using digital technology. — An electronic and manual search was conducted in the PubMed, Scopus, and Google Scholar databases. Publications of case reports and series written in English without data restrictions

SUMMARY:
Atrophied jaw is a condition where there is insufficient bone quantity to place root form implants. Several treatment plans are available for treating atrophied jaws, including subperiosteal implants. Subperiosteal implants were introduced in the last century. Poor clinical results led those implants to be progressively abandoned. Recently, several Authors suggested a revival of subperiosteal implants as an alternative to regenerative procedures.

DETAILED DESCRIPTION:
An electronic and manual search was conducted in the PubMed, Scopus, and Google Scholar databases. Publications of case reports and series written in English without data restrictions that reported on subperiosteal implants management of patients with severely atrophied jaws in completely and partially edentulous population.

The purpose of this systematic review of case reports and case series was to evaluate the spectrum of subperiosteal implants for severely atrophied jaws using digital technology.

ELIGIBILITY:
Inclusion Criteria:

* population with partial or fully edentulous arches, in particular Cawood and Howell class (IV-VI);

Exclusion Criteria:

* Articles were excluded if complex reconstructive surgery including bone grafts, barrier membranes, jaw osteotomies, sinus lift, alveolar ridge distraction, and zygomatic implants was recommended for treatment

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An electronic and manual search was conducted in the PubMed, Scopus, and Google Scholar databases. Publications of case reports and series written in English without data restrictions in the last 5 years.
Sampling Method: Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
to evaluate the spectrum of subperiosteal implants for severely atrophied jaws using digital technology. | 5 year retrospective
  The outcome was implant success or rejection.

SECONDARY OUTCOMES:
Biological complications | 5 year retrospective
  such as (dehiscence or exposure of the framework)

OTHER OUTCOMES:
Prosthetic complications | 5 year retrospective
  such as (fracture of the definitive or temporary prosthesis)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed ELSawy, PhD, Principal Investigator — Mansoura University
Locations (1):
- Mohammed El Sawy, Multiple Locations, Egypt

IPD SHARING:
Plan to Share IPD: No
just by contacting the corresponding author